CLINICAL TRIAL: NCT05985473
Title: Real-time Artificial Intelligence-based Speech Enhancement Methods for Hearing Aid Improvement
Acronym: REFINED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-016; 2023-A00140-45 (Other: ID RCB)
Record Dates: First submitted 2023-05-22; First posted 2023-08-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Deafness Neurosensory
Keywords: Spectrum of auditory neuropathy; speech enhancement; intelligibility; denoising methods; hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Professionally active adults with a moderate hearing loss (Other)
  Interventions: Other: audiological measurements; Other: Objective and subjective audiological measurements; Other: Evaluation of the denoising methods REFINED

INTERVENTIONS:
Other: audiological measurements — audiological measurements
Other: Objective and subjective audiological measurements — Objective and subjective audiological measurements
Other: Evaluation of the denoising methods REFINED — Evaluation of the denoising methods REFINED

SUMMARY:
Individuals with Auditory Neuropathy Spectrum Disorders (ANSD) represent 1-10% of adults with hearing loss. These individuals have little or no benefit from current hearing aids because ANSD is a continuum of hearing impairments due to synaptic or neural dysfunction in the peripheral and central parts of the auditory pathways, which impairs temporal information processing without necessarily affecting auditory sensitivity. There is a need to find ad-hoc denoising methods, based on the expert knowledge of audiologists, to improve the noise comprehension performance of these patients. Implemented denoising methods, based on artificial intelligence, will also greatly benefit more standard hearing loss cases.

DETAILED DESCRIPTION:
Longitudinal study consisting of multiple visits with multiple examinations over a total duration of approximately 3 years per ANSD participant and 1 year per normal hearing participant.

* normal hearing participant : year 1 : Inclusion visit, Phenotyping visit (Audiological tests), Follow-up Visit 1 (Noise Comprehension Tests)
* ANSD participant : year 1 : Inclusion visit, Phenotyping visit (Audiological tests), Follow-up Visit 1 (Noise Comprehension Tests) year 2 : Follow-up Visit 2 (Noise Comprehension Tests) year 3 : Follow-up Visit 3 (Noise Comprehension Tests)

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Age greater than or equal to 18 years,
* French mother tongue,
* Have an average tonal hearing loss (calculated according to the BIAP method) < 30 dB HL, on headphones, for each ear,
* Be professionally active, not be pre-retired and not be unemployed
* Be affiliated with a social security plan,

For participants with TSNA:

- Have degraded comprehension in noise (threshold of Intelligibility in Noise > 3 dB compared to the norm).

For controls:

- Have normal comprehension in noise (Intelligibility in Noise threshold ≤ 3 dB from the norm).

Exclusion Criteria:

For all participants:

* Have a conductive or mixed hearing loss, which is when the hearing loss affects both the outer and/or middle ear and the inner ear.
* Have an asymmetric hearing loss, i.e. a difference in average hearing loss between the left and right ear greater than 30 dB,
* Have sequelae of ear infections and/or a history of ENT disease that permanently affects hearing (vestibular schwannoma, Meniere's disease, sudden or fluctuating deafness, congenital hypoacusis)
* Being under guardianship,
* Being deprived of liberty by judicial or administrative decision, or being subject to legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of percentage of words correctly repeated by participants (ANSD and controls) | 3 years
  Evaluate intelligibility, i.e. the percentage of words correctly repeated, for different speech and noise conditions. Tests will be repeated with and without application of speech enhancement methods to the sound.

SECONDARY OUTCOMES:
Auditory Brain Response (ABRs) | 3 years
  Electrical activity of auditoral pathways, from the auditory nerve to the brain, in response to sound stimuli.
Percentage of words correctly repeated by participants with different angles of separation of speech and noises sources | 3 years
  Evaluate intelligibility and performance of source localisation for different angles of separation of speech and noises sources
Percentage of phonemes correctly repeated by participants (Verbo-Frequential Audiometry in the presence of calibrated noise: the DODELE AVfB test) | 3 years
  Evaluate speech perception in noise with phonemes as testing speech
Percentage of words correctly repeated by participants at different sound level of noise | 3 years
  Assess intelligibility in noise. Vocal tests will be repeated with and without tactile cues.
Myogenic vestibular evoked potentials (cervical VEMP or c-VEMP). | 3 years
  c-VEMP assesses the vestibular function through saccular and inferior vestibular nerve function performances. The collected parameters of c-VEMP testing include c-VEMP threshold, the latencies of the initial positivity (p1) and negativity (n1), and the p1-n1 inter-amplitude. We will collect these parameters and assess differences in controls vs. ANSDs.
Subjective evaluation of listening comfort using a visual analog scale | 3 years
  This self-assessment involves placing a cursor on a scale ranging from "very uncomfortable to very comfortable" using a scale ranging from 0 to 10.
Subjective evaluation of listening efficiency using a visual analog scale | 3 years
  This self-assessment involves placing a cursor on a scale ranging from "very inefficient to very efficient" using a scale ranging from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Avan, MD, Principal Investigator — CEntre de Recherche et d'Innovation en Audiologie Humain
Locations (1):
- CEntre de Recherche et d'Innovation en Audiologie Humaine, Paris, France